CLINICAL TRIAL: NCT02209038
Title: A Randomized Trial of Expanded Choice Sets to Increase Completion of Advance Directives
Brief Title: Choice Sets for Advance Directives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 820002
Record Dates: First submitted 2014-07-16; First posted 2014-08-05 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: End Stage Renal Disease
Keywords: end stage renal disease; hemodialysis; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Expanded AD Choice (Experimental): "Would you like to complete an advance directive with the assistance of any person(s) you choose?"
  4 answer choices:
  * Yes, I would like to complete a comprehensive version of an advance directive.
  * Yes, I would like to complete an expanded version of an advance directive.
  * Yes, I would like to complete a brief version of an advance directive.
  * No, I do not wish to complete an advance directive.
  Interventions: Behavioral: Expanded AD Choice
- Standard AD Choice (No Intervention): "Would you like to complete an advance directive with the assistance of any person(s) you choose?"
  2 answer choices:
  * Yes, I would like to complete an AD.
  * No, I do not wish to complete an advance directive.
- Expanded Life-sustaining therapy Choice (Experimental): For each hypothetical illness state described in the living will:
  4 answer choices:
  * No, I would not want life support.
  * Yes, I would want life support.
  * I would want life support if my doctor believes it could help, but I want to stop receiving life support if at any time my doctor believes it is only delaying the moment of my death.
  * I do not wish to specify a preference at this time.
  Interventions: Behavioral: Expanded Life-sustaining Therapy Choice
- Standard Life-sustaining Therapy Choice (No Intervention): For each hypothetical illness state described in the living will:
  3 answer choices:
  * No, I would not want life support.
  * Yes, I would want life support.
  * I do not wish to specify a preference at this time.

INTERVENTIONS:
Behavioral: Expanded AD Choice
  Arms: Expanded AD Choice
Behavioral: Expanded Life-sustaining Therapy Choice
  Arms: Expanded Life-sustaining therapy Choice

SUMMARY:
There is a large gap between the care seriously ill patients want and the care they receive. Advance directives (ADs) offer an opportunity for patients to express specific end-of-life preferences to avoid unwanted care. As promising as ADs may be for improving the quality of care near the end of life, rates of AD completion remain low and previous efforts to encourage their completion have had limited success. Principles of behavioral economics, such as the effects of defaults and other framing effects, may offer a novel approach to bridge the gap in end-of-life care. The goal of this study is to test whether the framing effect of expanding choice sets can increase the completion of and specification of choices within advance directives.

DETAILED DESCRIPTION:
This study has been designed as two sequential randomized trials to test two separate expanded choice set interventions, with the second randomization enrollment being contingent on results from the first. All enrolled subjects will be asked if they would like to complete an advance directive and will have been randomized to receive either an expanded answer choice set or a standard answer choice, as described in detail elsewhere. Only those subjects who express a desire to complete an advance directive from both arms will then be randomized again in a stratified fashion to receive either a standard advance directive or one with an expanded choice set for the decisions regarding life-sustaining therapy, as described in detail elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Proficient in English
* Chronic hemodialysis for minimum 90 days
* Does not currently have a living will

Exclusion Criteria:

* Blindness
* Cognitive impairment that prohibits subject's provision of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
advance directive | up to 4 weeks
  return of a completed and signed advance directive

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form-12v2 | baseline and 3 months
  change from baseline in Short Form-12v2 score at 3 months
McGill Quality of Life Questionnaire | baseline and 3 months
  change from baseline in McGill Quality of Life Questionnaire at 3 months
Satisfaction with Decision Scale | baseline
  satisfaction with decision scale measured at baseline after decision to complete an advance directive is made
Decisional Conflict Scale | up to 4 weeks
  Decisional Conflict Scale measured immediately after completion of an advance directive
no life-sustaining therapy preference specified | up to 4 weeks
  among all patients who complete an AD, the proportion of subjects who choose not to specify a preference for life-sustaining therapy on at least 1 clinical scenario within the AD

OTHER OUTCOMES:
hospital admissions | up to 4 years
  number of hospital admissions from enrollment to study completion
ICU admissions | up to 4 years
  number of ICU admissions from enrollment to study completion
Hospice admission | up to 4 years
death | up to 4 years
demographics of patients (ineligible) whom already completed a living will | enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, MD, PhD, Principal Investigator — University of Pennsylvania; Katherine R Courtright, MD, Study Director — University of Pennsylvania
Locations (15):
- United States (15):
  - Lourdes-Camden, Camden, New Jersey
  - Market Street DaVita, Philadelphia, Pennsylvania
  - Philadelphia 42nd Street DaVita, Philadelphia, Pennsylvania
  - Philadelphia PMC-Lombard DaVita, Philadelphia, Pennsylvania
  - University City DaVita, Philadelphia, Pennsylvania
  - Franklin DaVita, Philadelphia, Pennsylvania
  - PDI Walnut Tower DaVita, Philadelphia, Pennsylvania
  - Callowhill DaVita, Philadelphia, Pennsylvania
  - City Line DaVita, Philadelphia, Pennsylvania
  - South Broad Street, Philadelphia, Pennsylvania
  - Cottman DaVita, Philadelphia, Pennsylvania
  - South Philadelphia DaVita, Philadelphia, Pennsylvania
  - Radnor DaVita, Radnor, Pennsylvania
  - Abington DaVita, Willow Grove, Pennsylvania
  - Willow Grove DaVita, Willow Grove, Pennsylvania

REFERENCES:
- [Derived] Courtright KR, Madden V, Gabler NB, Cooney E, Kim J, Herbst N, Burgoon L, Whealdon J, Dember LM, Halpern SD. A Randomized Trial of Expanding Choice Sets to Motivate Advance Directive Completion. Med Decis Making. 2017 Jul;37(5):544-554. doi: 10.1177/0272989X16663709. Epub 2016 Aug 10. PMID 27510741